CLINICAL TRIAL: NCT05322538
Title: Menier's Disease - Bone Density Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Paker Miki, Attending physician, Otolaryngology head and neck surgery department, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EMC-22-0031
Record Dates: First submitted 2022-03-16; First posted 2022-04-12 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Meniere Disease; Osteoporosis; Osteopenia; Vitamin D Deficiency; Vestibular Disorder
MeSH Terms: conditions — Meniere Disease; Osteoporosis; Bone Diseases, Metabolic; Vitamin D Deficiency; Vestibular Diseases | interventions — Hearing Tests; Absorptiometry, Photon; Vestibular Evoked Myogenic Potentials; Audiometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (Other): Healthy controls with no known vestibular disease
  Interventions: Diagnostic Test: vitamin D plasma levels baseline; Diagnostic Test: Dual-energy X-ray absorptiometry at baseline; Diagnostic Test: Measuring Orthostatic Blood Pressure at baseline; Diagnostic Test: cold pressor test at baseline
- Definite Meniere's disease (Experimental): Patients with Definite Meniere's disease
  Interventions: Diagnostic Test: vitamin D plasma levels baseline; Diagnostic Test: Dual-energy X-ray absorptiometry at baseline; Diagnostic Test: cervical Vestibular evoked myogenic potentials at baseline; Diagnostic Test: Audiogram at baseline; Diagnostic Test: Measuring Orthostatic Blood Pressure at baseline; Diagnostic Test: cold pressor test at baseline; Diagnostic Test: vitamin D plasma levels one year after recruitment; Diagnostic Test: vitamin D plasma levels two years after recruitment; Diagnostic Test: Dual-energy X-ray absorptiometry one year after recruitment; Diagnostic Test: Dual-energy X-ray absorptiometry two years after recruitment; Diagnostic Test: cervical Vestibular evoked myogenic potentials one year after recruitment; Diagnostic Test: cervical Vestibular evoked myogenic potentials two years after recruitment; Diagnostic Test: Audiogram one year after recruitment; Diagnostic Test: Audiogram two years after recruitment; Diagnostic Test: Measuring Orthostatic Blood Pressure one year after recruitment; Diagnostic Test: Measuring Orthostatic Blood Pressure two years after recruitment; Diagnostic Test: cold pressor test one year after recruitment; Diagnostic Test: cold pressor test two years after recruitment

INTERVENTIONS:
Diagnostic Test: vitamin D plasma levels baseline — Measuring vitamin D plasma levels at baseline
Diagnostic Test: Dual-energy X-ray absorptiometry at baseline — Measuring T-score and Z-score of the femur and lumbar spine at baseline
  Other Names: DEXA
Diagnostic Test: cervical Vestibular evoked myogenic potentials at baseline — cVEMP is a vestibular test for saccular function, an otolith organ in the inner ear. the electrical response of the stermocledomastoid muscle to saccular stimulation is measured via two distinct waves - P13 and N23. the latency, amplitude and peak to peak amplitude will be measured.
  Other Names: cVEMP
  Arms: Definite Meniere's disease
Diagnostic Test: Audiogram at baseline — hearing measurement will be performed. Hearing level in dB will be performed in the 250-8,000 Hz frequency. The test includes Speech reception threshold and word recognition score.
  Other Names: Hearing test
  Arms: Definite Meniere's disease
Diagnostic Test: Measuring Orthostatic Blood Pressure at baseline — blood pressure will be measure two minutes after lying supine and repeated 3 minutes after standing. A drop of at least 20mmHg systolic pressure or at least 10mmHg diastolic blood pressure is considered a positive test
  Other Names: Orthostatic Hypotension
Diagnostic Test: cold pressor test at baseline — The cold pressor test is an indicator for sympathetic system function. A rise of at least 15mmHg of systolic pressure after putting the subject's hand in cold water (4 deg Celsius) is indicative of normal sympathetic function.
Diagnostic Test: vitamin D plasma levels one year after recruitment — Measuring vitamin D plasma levels one year after recruitment
  Arms: Definite Meniere's disease
Diagnostic Test: vitamin D plasma levels two years after recruitment — Measuring vitamin D plasma levels two years after recruitment
  Arms: Definite Meniere's disease
Diagnostic Test: Dual-energy X-ray absorptiometry one year after recruitment — Measuring T-score and Z-score of the femur and lumbar spine one year after recruitment
  Other Names: DEXA
  Arms: Definite Meniere's disease
Diagnostic Test: Dual-energy X-ray absorptiometry two years after recruitment — Measuring T-score and Z-score of the femur and lumbar spine two years after recruitment
  Arms: Definite Meniere's disease
Diagnostic Test: cervical Vestibular evoked myogenic potentials one year after recruitment — cVEMP is a vestibular test for saccular function, an otolith organ in the inner ear. the electrical response of the stermocledomastoid muscle to saccular stimulation is measured via two distinct waves - P13 and N23. the latency, amplitude and peak to peak amplitude will be measured one year after recruitment
  Other Names: cVEMP
  Arms: Definite Meniere's disease
Diagnostic Test: cervical Vestibular evoked myogenic potentials two years after recruitment — cVEMP is a vestibular test for saccular function, an otolith organ in the inner ear. the electrical response of the stermocledomastoid muscle to saccular stimulation is measured via two distinct waves - P13 and N23. the latency, amplitude and peak to peak amplitude will be measured two years after recruitment
  Other Names: cVEMP
  Arms: Definite Meniere's disease
Diagnostic Test: Audiogram one year after recruitment — hearing measurement will be performed. Hearing level in dB will be performed in the 250-8,000 Hz frequency. The test includes Speech reception threshold and word recognition score performed one year after recruitment
  Other Names: Hearing test
  Arms: Definite Meniere's disease
Diagnostic Test: Audiogram two years after recruitment — hearing measurement will be performed. Hearing level in dB will be performed in the 250-8,000 Hz frequency. The test includes Speech reception threshold and word recognition score performed two years after recruitment
  Other Names: Hearing test
  Arms: Definite Meniere's disease
Diagnostic Test: Measuring Orthostatic Blood Pressure one year after recruitment — blood pressure will be measure two minutes after lying supine and repeated 3 minutes after standing. A drop of at least 20mmHg systolic pressure or at least 10mmHg diastolic blood pressure is considered a positive test. The test will be performed one year after recruitment
  Other Names: Ortostatic hypostension
  Arms: Definite Meniere's disease
Diagnostic Test: Measuring Orthostatic Blood Pressure two years after recruitment — blood pressure will be measure two minutes after lying supine and repeated 3 minutes after standing. A drop of at least 20mmHg systolic pressure or at least 10mmHg diastolic blood pressure is considered a positive test. The test will be performed two year after recruitment.
  Other Names: Ostostatic hypotension
  Arms: Definite Meniere's disease
Diagnostic Test: cold pressor test one year after recruitment — The cold pressor test is an indicator for sympathetic system function. A rise of at least 15mmHg of systolic pressure after putting the subject's hand in cold water (4 deg Celsius) is indicative of normal sympathetic function. The test will be performed one year after recruitment.
  Arms: Definite Meniere's disease
Diagnostic Test: cold pressor test two years after recruitment — The cold pressor test is an indicator for sympathetic system function. A rise of at least 15mmHg of systolic pressure after putting the subject's hand in cold water (4 deg Celsius) is indicative of normal sympathetic function. The test will be performed two years after recruitment.
  Arms: Definite Meniere's disease

SUMMARY:
Meniere's disease is a progressive and debilitating inner ear disease characterised by vertigo and hearing loss. Several studies have linked Menierws disease with lower bone density and lower vitamin D levels. In the current prospective study definite Meniere's patients will be followed over a period of 2 year, during which repetitive measurements of bone density, vitamin D plasma levels, blood pressure as well as hearing and vestibular tests will be made. Results will be compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Definite Meniere's disease

Exclusion Criteria:

* hyperthyroidism
* hyperparathyroidism
* acromegaly
* hypogonadism
* diabetes melitus
* chronic renal failure
* alcoholism
* cushing syndrome
* rheumatoid arthritis
* systemic lupus erythematosus
* ankylosing spondylitis
* inflammatory bowel disease
* obstructive lung disease
* sarcoidosis
* amyloidosis
* celiac disease.
* chronic treatment with bisphosphonates
* chronic treatment with glucocorticoids
* chronic treatment with androgen deprivation therapy
* chronic treatment with gonadotropin releasing hormone agonist chronic treatment with aromatase inhibitor chronic treatment with loop diuretics chronic treatment with proton pump inhibitors chronic treatment with anti-seizure drugs chronic treatment with warfarin chronic treatment with SSRI chronic treatment with alpha or beta-blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin D plasma levels | baseline
  Vitamin D plasma levels
Vitamin D plasma levels | one year follow up
  Vitamin D plasma levels
Vitamin D plasma levels | two years follow-up
  Vitamin D plasma levels
Z-score and T-score of femur and lumbur spine | baseline
  DEXA exam - bone density. higher score means better resuls. osteopenia is defined as <-1 score , osteoporosis is defined as <-2.5 score
Z-score and T-score of femur and lumbur spine | one year follow up
  DEXA exam - bone density. higher score means better resuls. osteopenia is defined as <-1 score , osteoporosis is defined as <-2.5 score
Z-score and T-score of femur and lumbur spine | two years follow-up
  DEXA exam - bone density. higher score means better resuls. osteopenia is defined as <-1 score , osteoporosis is defined as <-2.5 score

SECONDARY OUTCOMES:
positive ortostatic hypotension | baseline
  drop of 20mmHg systolic blood pressure or drop of 10mmHG diastolic blood pressure after 3 minutes of standing up. all other results - negetive
positive ortostatic hypotension | one year follow up
  drop of 20mmHg systolic blood pressure or drop of 10mmHG diastolic blood pressure after 3 minutes of standing up. all other results - negetive
positive ortostatic hypotension | Two years follow-up
  drop of 20mmHg systolic blood pressure or drop of 10mmHG diastolic blood pressure after 3 minutes of standing up. all other results - negetive
cold pressure - autonomous sympatetic nervous system function - normal vs, inadequete | baseline
  a rise of less then 15mmHg after the test is considered inadequete function, more then 15hhHg - normal function
cold pressure - autonomous sympatetic nervous system function - normal vs, inadequete | one year follow up
  a rise of less then 15mmHg after the test is considered inadequete function, more then 15hhHg - normal function
cold pressure - autonomous sympatetic nervous system function - normal vs, inadequete | two years follow-up
  a rise of less then 15mmHg after the test is considered inadequete function, more then 15hhHg - normal function
ampitude, latency and peak to peak amplitude of the P13 and N23 waves in the cVEMP test | baseline
  cervical vestibular evoked myogenic potential exam
ampitude, latency and peak to peak amplitude of the P13 and N23 waves in the cVEMP test | one year follow up
  cervical vestibular evoked myogenic potential exam
ampitude, latency and peak to peak amplitude of the P13 and N23 waves in the cVEMP test | two years follow-up
  cervical vestibular evoked myogenic potential exam
Hearing level (dB), SRT in dB , descrimination in (%) in the audiology exam | baseline
  audiology exam
Hearing level (dB), SRT in dB , descrimination in (%) in the audiology exam | one year follow up
  audiology exam
Hearing level (dB), SRT in dB , descrimination in (%) in the audiology exam | two years follow-up
  audiology exam

IPD SHARING:
Plan to Share IPD: No